CLINICAL TRIAL: NCT00462085
Title: Muscle Activity With the Use of Ankle Foot Orthoses in Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: University Children's Hospital Basel (Other)
Other Study IDs: 94/04
Record Dates: First submitted 2007-04-17; First posted 2007-04-18 (Estimated); Last update posted 2007-04-18 (Estimated); Status verified 2007-04

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; ankle foot orthosis; emg; surface electromyography; gait analysis
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to investigate the change in muscle activity during gait with the use of ankle foot orthoses in children diagnosed with hemiplegic cerebral palsy.

DETAILED DESCRIPTION:
A small group of children with hemiplegic cerebral palsy is investigated by 3D instrumented gait analysis. Muscle activity is measured by surface electromyography (sEMG) of selected lower limb muscle groups. Kinematic, Kinetic, and sEMG data are compared between both lower limbs walking with and without an ankle foot orthosis. Data are also compared with those of an healthy control group.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of spastic hemiplegic cerebral palsy
* age between 8 and 18 years
* must have an equinus barefoot gait pattern
* must have a heel-toe gait pattern with ankle foot orthosis
* no prior operations

Exclusion Criteria:

* no Botulinumtoxin treatment for at least 6 months prior to investigation

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24
Dates: Start 2004-09; Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reinald Brunner, Prof.Dr.med., Study Director — University Children's Hospital Basel; Jacqueline Romkes, M.Sc., Principal Investigator — University Children's Hospital Basel
Locations (1):
- Laboratory for Movement Analysis, Basel, Canton of Basel-City, Switzerland